CLINICAL TRIAL: NCT06066021
Title: Evaluation of a Health Education Program for Type 2 Diabetes Patients
Acronym: EDUCA-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CEC/013/23
Record Dates: First submitted 2023-09-12; First posted 2023-10-04 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Retinopathy, Diabetic
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health education sessions for type 2 diabetic patients (Other): Patients will be pre-selected according to their risk of developing DR. It will be done through the Retina Risk® application. Will be invited to participate and followed. Retrospective and prospective data will be collected on medical and ophthalmological history (HbA1c value, if performed. 3 questionnaires will be carried out: DM disease, self-care, and emotional state, before and after awareness intervention about self-care through educational sessions in areas of greatest need (physical activity, nutrition, mental health, and self-care). The impact of the previously described sessions on the patients' health status will be assessed using 2 methods: By telephone and by physical examination. Repetition of the 3 questionnaires applied in V1.
  The Interventions will be made, through information sessions on the topics: mental health, nutrition, physical exercise, and care that diabetics must take to take care of their body.
  Interventions: Other: health educational sessions in diabetic patients type 2.

INTERVENTIONS:
Other: health educational sessions in diabetic patients type 2. — Professionals from different areas will be invited to carry out the sessions at Visit 2, namely on: mental health, physical activity, nutrition and self-care.

SUMMARY:
The goal of this, Retrospective and Prospective Low- Interventional study, is to implement health education interventions to promote self-care and reduce disease complications in DM Type 2 patients at higher risk of development/progression of Diabetic Retinopathy. ]. The main question it aims to answer are:

* To evaluate the impact of a health education intervention on mental health, self-care behaviors, and disease knowledge in patients with Diabetes Mellitus Type 2 with high risk of development/progression of Diabetic Retinopathy.
* To evaluate the impact of a health education intervention on the metabolic control of patients with Diabetes Mellitus Type 2 with high risk of development/progression of Diabetic Retinopathy.

Patients will have to (V1 and V4):

* answer three questionnaires, (Summary of Diabetes Self-Care Activities - SDSCA, QCD- Diabetes Knowledge Questionnaire and Depression Anxiety and Stress Scale" (DASS-21).
* measurement of weight and height, to calculate BMI.
* collection of glycated hemoglobin analysis (if they have been done in the last 3 months).

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is the most frequent complication of Diabetes mellitus and the main cause of legal blindness in working populations in industrialized countries.

A diagnosis of diabetes has important implications for individuals, not only for their health, but also because of the stigma that a diagnosis can bring, i.e., it can affect employment, quality of life, mental health, social opportunities, and other cultural aspects. These changes in the lives of diabetics can lead to stress. It is known that diabetes has a social and family connotation that leads to depression and anxiety appearing in parallel, which can influence the self-management that people must do in their daily lives. It is necessary to incorporate and integrate mental health care into all diabetic care.

Individuals with diabetes have difficulties: diagnosis, adherence to treatment, fear of complications and hypoglycemia, which can result in suffering, thus making self-management difficult.

In diabetic patients, the prevalence of symptoms of depression and anxiety is about two to four times higher than in the general population. Metabolic dysregulation influences brain function and disturbances in glucose regulation may be associated with depression. These emotions that arise can be disabling and very strong, leading the individual to often acquire behaviors that do not help in fighting the disease. There may be changes in eating behavior, or alcoholic beverages that are not favorable to glycemic control, that is, glycaemia rises proportionally to the most negative events in life, thus, stress leads to an increase in corticosteroids and consequently increases glycaemia. It is known that physical activity can reduce disease rates, namely diabetes, hypertension, obesity, among others. There are studies that show that physical activity is beneficial, whatever its intensity. It reduces the admission of chronically ill patients to hospitals, reduces pain and increases mental health and quality of life. With the development of physical activity programs applied to chronically ill patients, they are beneficial to promote the management of their disease, physical and mental health, and reduce the appearance of other comorbidities. In Diabetes Mellitus, the causes are complex, and its complications can be prevented with a healthy diet, normal blood glucose, adequate weight, and physical activity. For health professionals, who deal with these chronically ill patients, they have a huge challenge, since these people present risk behaviors (unhealthy eating and/or sedentary lifestyle). To assess the disease, there is glycosylated hemoglobin (HbA1c), which reflects the average blood glucose. It is used as a risk parameter and considered the gold standard for assessing glycemic control. The American Diabetes Association (ADA) sets HbA1c < 7% as the threshold of good control for most people with diabetes. To improve glycemic control, nutritional monitoring is important. Nutrition education is considered a preventive and treatment strategy to provide diabetic people with the necessary tools to face the change in lifestyle and achieve self-management of the disease. For this, it is necessary to increase knowledge, acquisition of skills, as well as promote the modification of attitudes and behaviors. It is important to increase people's active participation in the control and treatment of their disease.

Diabetics should participate in self-care education actions with the body, to improve the knowledge, skills, and abilities necessary for the self-care of this pathology.

Based on the evidence collected at the EYEMARKER (NCT02500862), CEC/009/17 study "Characterization of potential biomarkers of Eye Disease and Vision Loss", (ongoing at AIBILI), and STAR screening program "Development of a Model for Advanced Screening for Timely Treatment of Age-Related Eye Diseases", CEC/008/16, it was observed from the beginning the existence of individuals with DM who need clarification and education about their condition and about the care and behaviors to adopt to have a better management of their disease and avoid possible complications. With this study, it is intended to identify, in EYEMARKER patients who also participate in the STAR screening program, which individuals with Diabetes Mellitus are at greater risk of progression/development of Diabetic Retinopathy (DR), to better direct health education plans to reduce disease complications. The identification of patients at higher risk, who will be the target of health promotion actions, will be done through the "RetinaRisk" mobile phone application. After this analysis, 27 individuals who are at greater risk will be chosen. Self-care, knowledge about Diabetes Mellitus disease, emotional state, and metabolic control will be evaluated, before and after the health education sessions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 DM participating in STAR (CEC/008/16) and EYEMARKER (CEC/009/17)
* Higher risk patients through the RetinaRisk ® app ≥ 3%
* Age ≥50 years
* Body mass index (IMC) ≥ 25;
* Glycated hemoglobin (HbA1C): ≥6.5%; (7)
* Arterial hypertension (HTA): ≥ 139-89 (8)
* Presence of mild to moderate NPDR with presence of visible retina lesions (microaneurysms, hemorrhages, hard exudates and soft exudates)
* Subjects capable of understanding the information about the study and giving their informed consent to enter the study.
* Subjects willing and able to comply with the study.

Exclusion Criteria:

* Type 1 DM
* Moderately Severe NPDR;
* Presence of DME or PDR
* Other retinal vascular diseases than DR

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Change in Depression, Anxiety, and Stress Scale-21 (DASS-21) | 3 months
  total and subscales scores (depression; anxiety; stress) three months after the health education intervention training sessions. The scale score,(lower scores mean a better result), (the minimum and maximum values): 0 - Nothing applied to me
  1. - It applied to me a few times
  2. - It has applied to me many times
  3. - It applied to me most of the time
Change in the Summary of Diabetes Self-Care Activities (SDSCA) | 3 months
  total and subscales scores (general diet; specific diet; exercise; blood-glucose testing; foot-care; smoking) three months after the health education intervention training sessions.
  The scale used is number of days (from 0 to 7)
Change in the Diabetes Knowledge Questionnaire (DKQ - Portuguese version) | 3 months
  Subscales scores (treatment, control and complications; causes; duration) three months after the health education intervention training sessions.
  This consists of 20 items distributed by three dimensions (Treatment, control and complications, Causes and Duration).The minimum and maximum values is 0-100, the 0 is minimum and 100 is maximum

SECONDARY OUTCOMES:
Measure the change in the blood HbA1C level | 3 months
  Measure the change in the blood HbA1C level after the health education intervention training sessions.
  The unit of measurement for HbA1c is in percentage (%).
Measure the change in BMI | 3 months
  Measure the change in BMI after the health education intervention training sessions.
  The unit of measurement for BMI is expressed in units of kg/m2 (weight in kilograms and height in meters).

CONTACTS AND LOCATIONS:
Locations (1):
- AIBILI-CEC (AIBILI- Clinical Trials Centre), Coimbra, Portugal

REFERENCES:
- [Background] Eisma JH, Dulle JE, Fort PE. Current knowledge on diabetic retinopathy from human donor tissues. World J Diabetes. 2015 Mar 15;6(2):312-20. doi: 10.4239/wjd.v6.i2.312. PMID 25789112
- [Background] Ambury T. Mental health in diabetes: can't afford to address the service gaps or can't afford not to? Br J Gen Pract. 2020 Feb 27;70(692):108-109. doi: 10.3399/bjgp20X708365. Print 2020 Mar. No abstract available. PMID 32107219
- [Background] Kozlowska O, Solomons L, Cuzner D, Ahmed S, McManners J, Tan GD, Lumb A, Rea R. Diabetes care: closing the gap between mental and physical health in primary care. Br J Gen Pract. 2017 Oct;67(663):471-472. doi: 10.3399/bjgp17X692993. No abstract available. PMID 28963429
- [Background] Alessi J, de Oliveira GB, Franco DW, Brino do Amaral B, Becker AS, Knijnik CP, Kobe GL, de Carvalho TR, Telo GH, Schaan BD, Telo GH. Mental health in the era of COVID-19: prevalence of psychiatric disorders in a cohort of patients with type 1 and type 2 diabetes during the social distancing. Diabetol Metab Syndr. 2020 Aug 31;12:76. doi: 10.1186/s13098-020-00584-6. eCollection 2020. PMID 32879637
- [Background] Cheval B, Finckh A, Maltagliati S, Fessler L, Cullati S, Sander D, Friese M, Wiers RW, Boisgontier MP, Courvoisier DS, Luthy C. Cognitive-bias modification intervention to improve physical activity in patients following a rehabilitation programme: protocol for the randomised controlled IMPACT trial. BMJ Open. 2021 Sep 21;11(9):e053845. doi: 10.1136/bmjopen-2021-053845. PMID 34548372
- [Background] Funnell MM, Brown TL, Childs BP, Haas LB, Hosey GM, Jensen B, Maryniuk M, Peyrot M, Piette JD, Reader D, Siminerio LM, Weinger K, Weiss MA. National standards for diabetes self-management education. Diabetes Care. 2009 Jan;32 Suppl 1(Suppl 1):S87-94. doi: 10.2337/dc09-S087. No abstract available. PMID 19118294
- [Background] Use of Glycated Haemoglobin (HbA1c) in the Diagnosis of Diabetes Mellitus: Abbreviated Report of a WHO Consultation. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK304267/ PMID 26158184
- [Background] Sociedade Portuguesa de Hipertensão. (2020). Sociedade Portuguesa de Hipertensão. Sociedade Portuguesa de Hipertensão. https://www.sphta.org.pt/pt/base8_detail/24/89
- [Background] Ebrahem, S. M., & Masry, S. E. (2017). Effect of relaxation therapy on depression, anxiety, stress and quality of life among diabetic patients. Clinical Nursing Studies, 5(1), 35. https://doi.org/10.5430/cns.v5n1p35
- [Background] Trief PM, Izquierdo R, Eimicke JP, Teresi JA, Goland R, Palmas W, Shea S, Weinstock RS. Adherence to diabetes self care for white, African-American and Hispanic American telemedicine participants: 5 year results from the IDEATel project. Ethn Health. 2013;18(1):83-96. doi: 10.1080/13557858.2012.700915. Epub 2012 Jul 5. PMID 22762449
- [Background] Sousa, M. R., Pereira, F., Martins, T., Rua, I., Ribeiro, I., Cerdeira, C., Lopes, L., Sèvegrand, C., & Santos, C. (2019). Impact of an educational programme in Portuguese people with diabetes. Action Research, 17(2), 258-276. https://doi.org/10.1177/1476750317736369